CLINICAL TRIAL: NCT06030843
Title: The Treatment Effects of Empagliflozin on Renal Outcomes in Cardiorenal Syndrome Type 1
Acronym: TREAT-CRS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 674/66
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Empagliflozin in Cardiorenal Syndrome Type 1
Keywords: Empagliflozin; SGLT2i; Cardiorenal syndrome; ADHF; AKI
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empagliflozin (Experimental): Empagliflozin 10 mg po OD
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Empagliflozin 10 MG
  Arms: Empagliflozin
Drug: Placebo — Matching placebo containing Lactose content (0.26 gram)
  Arms: Placebo

SUMMARY:
Effects of Empagliflozin compared with placebo in cardiorenal syndrome type 1, evaluated by MAKE30.

ELIGIBILITY:
Inclusion criteria

* Age 18 years or more
* Hospitalized for the primary diagnosis of acute denovo or decompensated chronic heart regardless of ejection fraction
* AKI KDIGO any stage or urine NGAL ≥ 150 ng/mL
* Must be able to be enrolled into the trial ≤ 12 hours of diagnosis of AKI or elevated urine NGAL

Exclusion criteria

* Denied to participate in the study
* Cardiogenic shock or unstable hemodynamic (systolic blood pressure of at least 100 mmHg or required inotropic support within last 24 hours)
* Cardiac mechanical support (i.e. extracorporeal membrane oxygenation and intra-aortic balloon pump)
* Acute coronary syndrome
* Diagnosed with cause of AKI other than cardiorenal syndrome (eg. sepsis, nephrotoxic, dehydration)
* Anuria or requiring dialysis or expected to required dialysis within 24 hr
* Baseline eGFR ≤ 20 ml/min/1.73m2 with or without dialysis initiated
* Heart or kidney transplanted
* Previously received any SGLT2i in the last 3 months before admission
* Allergic to any SGLT2i
* Type 1 diabetes mellitus
* History of ketoacidosis, including diabetic ketoacidosis
* Pregnancy
* Comorbid conditions with an expected survival of less than 1 months such as end-stage liver or heart disease, or uncurable malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MAKE30 | 30 days
  The composite outcome of death, new dialysis, and sustained loss of kidney function (which was defined as a 25% or greater decline in eGFR from baseline) assess at 30 days following randomization

SECONDARY OUTCOMES:
In-hospital mortality rate | During admission
  In-hospital mortality rate
30-days mortality rate | 30 days
  30-days mortality rate
Initiation of Renal Replacement therapy | 30 days
  Initiation of Renal Replacement therapy
Sustained loss of kidney function defined as a 25% or greater decline in eGFR at 30 days following randomisation compared to baseline eGFR | 30 days
  Sustained loss of kidney function defined as a 25% or greater decline in eGFR at 30 days following randomisation compared to baseline eGFR
Recurrent heart failure | 30 days
  Recurrent heart failure required hospital administration
Vasoactive drug | 30 days
  Vasoactive drug use
Mechanical ventilation | 30 days
  Mechanical ventilation use
Ventricular tachycardia or ventricular fibrillation | 30 days
  Ventricular tachycardia or ventricular fibrillation
Resuscitation following a cardiac arrest | 30 days
  Resuscitation following a cardiac arrest
Reduction of prespecified renal biomarkers | 30 days
  Reduction of prespecified renal biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Nattachai Srisawat, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Pathumwan, Thailand

IPD SHARING:
Plan to Share IPD: Undecided